CLINICAL TRIAL: NCT05609396
Title: Interventions to Improve Bowel Cancer Screening Uptake in Ireland: a 2x2 Factorial Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dublin City University (Other)
Collaborators: The National Screening Service (Unknown); Newcastle University (Other); University College, London (Other); University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Nicholas Clarke, Principal Investigator, Dublin City University
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: BSA_012
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; Fecal Immunochemical test; cancer screening; Uptake; Participation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a 2x2 factorial design non-randomised control trial. This design will test main effects of each intervention and investigate whether the two interventions interact (25). Individuals between the ages of 60-62 (new invitees) will be sampled from invitees who do not respond to the initial screening invitation and allocated to one of four trial arms using batch randomisation. The four trial arms will be:
  1. Usual care - Standard reminder and no test kit
  2. Standard reminder plus test kit
  3. Theoretically informed behavioural intervention (modified reminder letter) at reminder and no test kit
  4. Theoretically informed behavioural intervention at reminder with test kit The main effect of the test kit is estimated by comparing 2+4 vs 1+3; main effect of behavioural intervention is estimated from 3+4 vs 1+2.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual care (No Intervention): Standard reminder letter only
- Enhanced reminder letter only (Experimental): Behaviorally enhanced reminder letter
  Interventions: Behavioral: Behaviorally enhanced reminder letter
- Usual care plus test kit (Experimental): Standard reminder letter plus test kit
  Interventions: Behavioral: Behaviorally enhanced reminder letter
- Enhanced reminder plus test kit (Experimental): Behaviorally enhanced reminder letter plus test kit
  Interventions: Behavioral: Behaviorally enhanced reminder letter

INTERVENTIONS:
Behavioral: Behaviorally enhanced reminder letter — Behavioral interventions to increase FIT-based colorectal cancer screening uptake
  Other Names: Direct mailing of FIT test kit; Behaviorally enhanced reminder letter and direct mailing of FIT kit
  Arms: Enhanced reminder letter only; Enhanced reminder plus test kit; Usual care plus test kit

SUMMARY:
High uptake is vital to population-based screening. BowelScreen (Irelands national organised population-based colorectal cancer screening programme) has not achieved recommended screening uptake targets. In Ireland sending the test kit in the screening invitation reminder may be an important strategy in targeting non-responders and would address a key difference between Ireland and other international screening programmes with higher uptake. In addition, few studies have focused on behavioural barriers to screening participation. Founded upon the MRC Guidelines for the Development of Complex Interventions, our systematic, theoretically-informed investigation of FIT screening participation has begun to identify behavioural antecedents to screening participation in Ireland. This study will implement a multilevel evidence-based, theoretically-informed intervention which includes the automatic inclusion of the test kit in the screening reminder, alone and in combination with an intervention to influence individuals' screening participation. This multilevel intervention will provide recommendations for the screening invitation delivery, potentially bringing the programme closer to recommended uptake targets (50%) and in the long-term influence reductions in bowel cancer incidence and mortality in Ireland.

DETAILED DESCRIPTION:
To achieve population-level health gains, colorectal cancer screening programmes require high uptake. Guidelines recommend uptake of 65%-75%. In Ireland, faecal immunochemical test (FIT)-based screening uptake is considerably lower than this (around 40%), despite FIT being recommended as the screening test of choice given its potential to deliver higher uptake than other tests. As well as being suboptimal overall, uptake in Ireland is significantly lower among males and lower socioeconomic groups the very groups at higher underlying risk of colorectal cancer. While improving overall uptake is important, focus is also needed on reducing differentials in uptake; left unchecked these may lead to further disparities in health outcomes among those most at risk.

The main difference between Ireland's screening programme and programmes with higher uptake is that BowelScreen does not send the test kit with the screening invitation: invitees are required to contact a call-centre, consent to participate and request the kit. Uptake in Ireland is 10-30% lower than Scotland, the Netherlands and England and, indeed, in a pilot screening programme in Dublin that also sent the test automatically.

Internationally, various strategies to improve uptake have been tested. Some studies report increases using advance notification letters, postal mailing of home-based testing kits, and telephone contacts but many studies have been negative. Recent UK research points to potential in intervening among non-responders to the initial screening invitation, but few intervention studies have focussed on non-responders. An important limitation of existing studies is that most investigators failed to base their interventions on an understanding of what influences individuals' decisions about screening participation/non-participation.

A range of barriers to uptake have been identified and include fatalism, poor knowledge, being poorly informed about cancer and screening and holding negative attitudes, beliefs and emotions towards FIT screening. Following the MRC Framework for the Development of Complex Interventions and being theoretically informed, this work has the explicit intention of informing future interventions.

This proposal seeks to test efficacy in increasing uptake of two interventions among non responders: 1) including a test kit with the current reminder, and 2) an evidence-based and theoretically informed behavioural intervention (e.g. modified reminder letter, modified accompanying leaflet).

ELIGIBILITY:
Inclusion Criteria:

All new invitees of Irelands National BowelScreen Programme Individuals aged 60-64

Exclusion Criteria:

All individuals who are within the screening age range of Irelands national bowel screening programme are eligible to be included.

Ages: 60 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8734 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Uptake | 3 months from intervention delivery
  Participation rate in each arm

SECONDARY OUTCOMES:
Uptake by deprivation, sex and age | 3 months from intervention delivery
  Participation rate in each arm by deprivation, sex and age

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Clarke, PhD, Principal Investigator — DCU
Locations (1):
- National Screening Service, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weller DP, Patnick J, McIntosh HM, Dietrich AJ. Uptake in cancer screening programmes. Lancet Oncol. 2009 Jul;10(7):693-9. doi: 10.1016/S1470-2045(09)70145-7. PMID 19573798
- [Background] Essink-Bot ML, Dekker E. Equal access to colorectal cancer screening. Lancet. 2016 Feb 20;387(10020):724-6. doi: 10.1016/S0140-6736(15)01221-0. Epub 2015 Dec 9. No abstract available. PMID 26680216
- [Background] European Colorectal Cancer Screening Guidelines Working Group; von Karsa L, Patnick J, Segnan N, Atkin W, Halloran S, Lansdorp-Vogelaar I, Malila N, Minozzi S, Moss S, Quirke P, Steele RJ, Vieth M, Aabakken L, Altenhofen L, Ancelle-Park R, Antoljak N, Anttila A, Armaroli P, Arrossi S, Austoker J, Banzi R, Bellisario C, Blom J, Brenner H, Bretthauer M, Camargo Cancela M, Costamagna G, Cuzick J, Dai M, Daniel J, Dekker E, Delicata N, Ducarroz S, Erfkamp H, Espinas JA, Faivre J, Faulds Wood L, Flugelman A, Frkovic-Grazio S, Geller B, Giordano L, Grazzini G, Green J, Hamashima C, Herrmann C, Hewitson P, Hoff G, Holten I, Jover R, Kaminski MF, Kuipers EJ, Kurtinaitis J, Lambert R, Launoy G, Lee W, Leicester R, Leja M, Lieberman D, Lignini T, Lucas E, Lynge E, Madai S, Marinho J, Maucec Zakotnik J, Minoli G, Monk C, Morais A, Muwonge R, Nadel M, Neamtiu L, Peris Tuser M, Pignone M, Pox C, Primic-Zakelj M, Psaila J, Rabeneck L, Ransohoff D, Rasmussen M, Regula J, Ren J, Rennert G, Rey J, Riddell RH, Risio M, Rodrigues V, Saito H, Sauvaget C, Scharpantgen A, Schmiegel W, Senore C, Siddiqi M, Sighoko D, Smith R, Smith S, Suchanek S, Suonio E, Tong W, Tornberg S, Van Cutsem E, Vignatelli L, Villain P, Voti L, Watanabe H, Watson J, Winawer S, Young G, Zaksas V, Zappa M, Valori R. European guidelines for quality assurance in colorectal cancer screening and diagnosis: overview and introduction to the full supplement publication. Endoscopy. 2013;45(1):51-9. doi: 10.1055/s-0032-1325997. Epub 2012 Dec 4. PMID 23212726
- [Background] BowelScreen. BowelScreen: Programme Statistical Bulletin 2016 - 2017 [Internet]. 2018 [cited 2019 Oct 29]. Available from: http://www.screeningservice.ie/publications/BowelScreen_statistical_bulletin_2016-2017_FINAL%203_7_19.pdf
- [Background] Allison JE, Fraser CG, Halloran SP, Young GP. Population screening for colorectal cancer means getting FIT: the past, present, and future of colorectal cancer screening using the fecal immunochemical test for hemoglobin (FIT). Gut Liver. 2014 Mar;8(2):117-30. doi: 10.5009/gnl.2014.8.2.117. Epub 2014 Mar 11. PMID 24672652
- [Background] Digby J, McDonald PJ, Strachan JA, Libby G, Steele RJ, Fraser CG. Use of a faecal immunochemical test narrows current gaps in uptake for sex, age and deprivation in a bowel cancer screening programme. J Med Screen. 2013 Jun;20(2):80-5. doi: 10.1177/0969141313497197. Epub 2013 Jul 18. PMID 24009088
- [Background] Vart G, Banzi R, Minozzi S. Comparing participation rates between immunochemical and guaiac faecal occult blood tests: a systematic review and meta-analysis. Prev Med. 2012 Aug;55(2):87-92. doi: 10.1016/j.ypmed.2012.05.006. Epub 2012 May 23. PMID 22634386
- [Background] Clarke N, Sharp L, Osborne A, Kearney PM. Comparison of uptake of colorectal cancer screening based on fecal immunochemical testing (FIT) in males and females: a systematic review and meta-analysis. Cancer Epidemiol Biomarkers Prev. 2015 Jan;24(1):39-47. doi: 10.1158/1055-9965.EPI-14-0774. Epub 2014 Nov 6. PMID 25378366
- [Background] Clarke N, McNamara D, Kearney PM, O'Morain CA, Shearer N, Sharp L. The role of area-level deprivation and gender in participation in population-based faecal immunochemical test (FIT) colorectal cancer screening. Prev Med. 2016 Dec;93:198-203. doi: 10.1016/j.ypmed.2016.10.012. Epub 2016 Oct 18. PMID 27765660
- [Background] Wardle J, Robb K, Vernon S, Waller J. Screening for prevention and early diagnosis of cancer. Am Psychol. 2015 Feb-Mar;70(2):119-33. doi: 10.1037/a0037357. PMID 25730719
- [Background] Clarke N, Sharp L, O'Leary E, Richardson N. A report on the excess burden of cancer among men in the Republic of Ireland. 2013 [cited 2015 Aug 14]; Available from: https://www.lenus.ie/hse/handle/10147/316719
- [Background] NHS Highland. DPH Annual Report 2019 and appendices [Internet]. Scotland; 2019 [cited 2020 Jan 17]. Available from: https://www.nhshighland.scot.nhs.uk/Publications/Documents/DPH-Annual-Report-2019-and-appendices.pdf
- [Background] Douma LN, Uiters E, Timmermans DR. The Dutch public are positive about the colorectal cancer-screening programme, but is this a well-informed opinion? BMC Public Health. 2016 Nov 29;16(1):1208. doi: 10.1186/s12889-016-3870-7. PMID 27899154
- [Background] Hirst Y, Stoffel S, Baio G, McGregor L, von Wagner C. Uptake of the English Bowel (Colorectal) Cancer Screening Programme: an update 5 years after the full roll-out. Eur J Cancer. 2018 Nov;103:267-273. doi: 10.1016/j.ejca.2018.07.135. Epub 2018 Sep 7. PMID 30196989
- [Background] McNamara D, Leen R, Seng-Lee C, Shearer N, Crotty P, Neary P, Walsh P, Boran G, O'Morain C. Sustained participation, colonoscopy uptake and adenoma detection rates over two rounds of the Tallaght-Trinity College colorectal cancer screening programme with the faecal immunological test. Eur J Gastroenterol Hepatol. 2014 Dec;26(12):1415-21. doi: 10.1097/MEG.0000000000000207. PMID 25244415
- [Background] Rat C, Latour C, Rousseau R, Gaultier A, Pogu C, Edwards A, Nguyen JM. Interventions to increase uptake of faecal tests for colorectal cancer screening: a systematic review. Eur J Cancer Prev. 2018 May;27(3):227-236. doi: 10.1097/CEJ.0000000000000344. PMID 28665812
- [Background] Issaka RB, Avila P, Whitaker E, Bent S, Somsouk M. Population health interventions to improve colorectal cancer screening by fecal immunochemical tests: A systematic review. Prev Med. 2019 Jan;118:113-121. doi: 10.1016/j.ypmed.2018.10.021. Epub 2018 Oct 24. PMID 30367972
- [Background] Sabatino SA, Lawrence B, Elder R, Mercer SL, Wilson KM, DeVinney B, Melillo S, Carvalho M, Taplin S, Bastani R, Rimer BK, Vernon SW, Melvin CL, Taylor V, Fernandez M, Glanz K; Community Preventive Services Task Force. Effectiveness of interventions to increase screening for breast, cervical, and colorectal cancers: nine updated systematic reviews for the guide to community preventive services. Am J Prev Med. 2012 Jul;43(1):97-118. doi: 10.1016/j.amepre.2012.04.009. PMID 22704754
- [Background] Wardle J, von Wagner C, Kralj-Hans I, Halloran SP, Smith SG, McGregor LM, Vart G, Howe R, Snowball J, Handley G, Logan RF, Rainbow S, Smith S, Thomas MC, Counsell N, Morris S, Duffy SW, Hackshaw A, Moss S, Atkin W, Raine R. Effects of evidence-based strategies to reduce the socioeconomic gradient of uptake in the English NHS Bowel Cancer Screening Programme (ASCEND): four cluster-randomised controlled trials. Lancet. 2016 Feb 20;387(10020):751-9. doi: 10.1016/S0140-6736(15)01154-X. Epub 2015 Dec 9. PMID 26680217
- [Background] Kerrison RS, McGregor LM, Marshall S, Isitt J, Counsell N, Wardle J, von Wagner C. Use of a 12 months' self-referral reminder to facilitate uptake of bowel scope (flexible sigmoidoscopy) screening in previous non-responders: a London-based feasibility study. Br J Cancer. 2016 Mar 29;114(7):751-8. doi: 10.1038/bjc.2016.43. Epub 2016 Mar 15. PMID 26977856
- [Background] Clarke N, Gallagher P, Kearney PM, McNamara D, Sharp L. Impact of gender on decisions to participate in faecal immunochemical test-based colorectal cancer screening: a qualitative study. Psychooncology. 2016 Dec;25(12):1456-1462. doi: 10.1002/pon.4085. Epub 2016 Feb 11. PMID 26864167
- [Background] Clarke N, Kearney PM, Gallagher P, McNamara D, O'Morain CA, Sharp L. Negative emotions and cancer fatalism are independently associated with uptake of Faecal Immunochemical Test-based colorectal cancer screening: Results from a population-based study. Prev Med. 2021 Apr;145:106430. doi: 10.1016/j.ypmed.2021.106430. Epub 2021 Jan 19. PMID 33482227
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Background] Cane J, O'Connor D, Michie S. Validation of the theoretical domains framework for use in behaviour change and implementation research. Implement Sci. 2012 Apr 24;7:37. doi: 10.1186/1748-5908-7-37. PMID 22530986